CLINICAL TRIAL: NCT02873663
Title: Biomarkers for the Detection of Heavy Alcohol Use in Patients With and Without Liver Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Diagnostic
Other Study IDs: S53031
Record Dates: First submitted 2011-04-13; First posted 2016-08-19 (Estimated); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Alcohol Abuse; Liver Disease
MeSH Terms: conditions — Alcoholism; Liver Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- heavy drinkers (Experimental): Plasma and head hair collection
  Interventions: Procedure: Plasma and head hair collection
- teetotalers (Experimental): Plasma and head hair collection
  Interventions: Procedure: Plasma and head hair collection

INTERVENTIONS:
Procedure: Plasma and head hair collection — Plasma and head hair collection

SUMMARY:
The investigators will test the validity of biomarkers for the detection of heavy alcohol use in patients with and without liver disease.

DETAILED DESCRIPTION:
The investigators will test the validity of biomarkers for the detection of heavy alcohol use in patients with and without liver disease.

The investigators will test the validity of carbohydrate deficient transferrin (CDT)(using capillary zone electrophoresis) in blood and ethyl glucuronide (EtG)(using Liquid Chromatography-MS-MS) in hair in patients with heavy alcohol use, moderate alcohol use and patients who do not drink alcohol.

ELIGIBILITY:
Inclusion Criteria:

* patients who do not drink alcohol, moderate drinkers (between 0 and 60 g a day) and patients who drink 60 or more grams alcohol a day

Exclusion criteria

* refusal for inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2010-12 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
level of disialotransferrin in blood (expressed as percentage di-sialotransferrin) and ethyl glucuronide (expressed in pg/mg) in hair | single determination at inclusion (both on the same day, when patient is seen at the outpatient clinic or when admitted to the hospital) without follow-up
  Blood and hair will be collected at one single time-point (procedure of blood and hair sampling takes 30 min) to measure serum CDT and hair ethylglucuronide levels (markers of alcohol use in the prior time period) when the patient presents itself at the hospital, without further follow-up.

SECONDARY OUTCOMES:
influence of the stage of liver and renal impairment on serum CDT and hair EtG | on the basis of a single determination which is done for the standard care (when patient is seen at the outpatient clinic or when admitted to the hospital)
  Blood and hair will be collected at one single time-point (procedure of blood and hair sampling takes 30 min) to measure serum CDT and hair ethylglucuronide levels (markers of alcohol use in the prior time period) when the patient presents itself at the hospital, without further follow-up. Liver and kidney parameters are analyzed in the blood in the context of standard care.

CONTACTS AND LOCATIONS:
Overall Officials: Jef Verbeek, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams Brabant, Belgium